CLINICAL TRIAL: NCT07240532
Title: Efficacy of a Multimodal Physiotherapy Program and Mobile-App Guided Meditation in Adults With Frequent or Chronic Tension-Type Headache: A Randomized Clinical Trial
Brief Title: Efficacy of a Multimodal Physiotherapy Program and Mobile-App Guided Meditation in Adults With Frequent or Chronic Tension-Type Headache
Acronym: JBE-CEF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Jihane Boudount El Kadaoui, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JBE-CEF-2025
Record Dates: First submitted 2025-11-16; First posted 2025-11-21 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Tension-Type Headache; Chronic Tension-type Headache; Frequent Episodic Tension-Type Headache
Keywords: Tension-Type Headache; Chronic Tension-Type Headache; Multimodal Physiotherapy; Manual Therapy; Dry Needling; Mindfulness; Guided Meditation; Mobile Application; Non-Pharmacological Treatment; Randomized Controlled Trial; Biopsychophysiological Approach;; Pain Management; Headache Disability
MeSH Terms: conditions — Tension-Type Headache; Agnosia | interventions — Musculoskeletal Manipulations; Dry Needling

STUDY DESIGN:
Intervention Model Description: This is a three-arm parallel randomized controlled trial with equal allocation (1:1:1). Participants will be randomly assigned to one of three groups: multimodal physiotherapy, guided meditation via mobile app, or combined treatment (physiotherapy plus meditation).
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded to their group assignment to minimize expectation bias. Outcome assessors will also be blinded to intervention allocation. Therapists and investigators will not be blinded due to the nature of the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Multimodal Physiotherapy (Experimental): Participants in this group will receive a multimodal physiotherapy program once a week for four weeks. Each session includes thoracic (T4-T7) and cervicothoracic (C7-T1) manipulation, suboccipital inhibition, deep dry needling of the upper trapezius and sternocleidomastoid muscles, specific massage (temporal, paracervical, and SCM muscles), and passive cervical mobilization in rotation and lateral flexion within a pain-free range.
  Interventions: Other: Multimodal Physiotherapy for Tension-Type Headache
- Guided Meditation Group (Experimental): Participants in this group will use the Insight Timer mobile application to perform daily guided meditation sessions lasting approximately 5-7 minutes, focused on mindfulness, stress reduction, and sleep improvement. Only free, Spanish-language content from the app will be used. The program will last four weeks.
  Interventions: Behavioral: Guided Meditation Using Insight Timer App
- Combined Multimodal Physiotherapy and Guided Meditation (Experimental): Participants in this group will receive both interventions: one weekly session of multimodal physiotherapy for four weeks and daily guided meditation using the Insight Timer app (approximately 5-7 minutes per day).
  Interventions: Other: Multimodal Physiotherapy for Tension-Type Headache; Behavioral: Guided Meditation Using Insight Timer App

INTERVENTIONS:
Other: Multimodal Physiotherapy for Tension-Type Headache — Participants in this group will receive a multimodal physiotherapy program once a week for four weeks. Each session includes thoracic (T4-T7) and cervicothoracic (C7-T1) manipulation, suboccipital inhibition, deep dry needling of the upper trapezius and sternocleidomastoid muscles, specific massage (temporal, paracervical, and SCM muscles), and passive cervical mobilization in rotation and lateral flexion within a pain-free range. All procedures will be performed by a physiotherapist with over ten years of clinical experience.
  Other Names: Physiotherapy Multimodal Program; Manual Therapy plus Dry Needling
  Arms: Combined Multimodal Physiotherapy and Guided Meditation; Multimodal Physiotherapy
Behavioral: Guided Meditation Using Insight Timer App — Participants in this group will use the Insight Timer mobile application to perform daily guided meditation sessions of approximately 5-7 minutes for four weeks. All sessions will use free Spanish-language content focused on mindfulness, stress reduction, and sleep improvement. Participants will receive written instructions to ensure adherence.
  Other Names: Mobile Mindfulness Meditation; Digital Mindfulness Training
  Arms: Combined Multimodal Physiotherapy and Guided Meditation; Guided Meditation Group

SUMMARY:
The goal of this clinical trial is to evaluate whether a multimodal physiotherapy program and guided meditation using a mobile app can help reduce headache pain and improve quality of life in adults with frequent or chronic tension-type headache. The study analyzes the effects of physical and psychological interventions applied both separately and in combination, so that the combined treatment addresses tension-type headache as a multifactorial condition influenced by biopsychophysiological factors, integrating physical and psychological strategies to improve participants' overall well-being.

The main questions it aims to answer are:

* Does multimodal physiotherapy lower the intensity and frequency of headaches?
* Does guided meditation through a mobile app help reduce stress and improve emotional well-being?
* Are the combined effects of physiotherapy and meditation greater than either intervention alone?

The study will compare:

* A group receiving multimodal physiotherapy sessions once a week for four weeks,
* A group practicing guided meditation with a mobile app for about 5 to 7 minutes daily,
* A group combining both physiotherapy and meditation.

Participants will:

* Attend clinical sessions or use the meditation app depending on group assignment,
* Complete short questionnaires about pain, stress, sleep, and daily functioning,
* Record headache episodes in a structured diary during the study period.

DETAILED DESCRIPTION:
Tension-type headache (TTH) is one of the most prevalent primary headache disorders and a major cause of pain-related disability worldwide. Its multifactorial nature involves musculoskeletal, psychological, and neurophysiological mechanisms, leading to recurrent episodes of pain and functional impairment. Conventional management often provides limited relief, highlighting the need for integrative, non-pharmacological approaches.

This randomized controlled clinical trial is designed to evaluate the efficacy of multimodal physiotherapy and guided meditation delivered through a mobile application, both separately and in combination, in adults with frequent or chronic TTH. The combined intervention is intended to address TTH as a multifactorial condition influenced by biopsychophysiological factors, integrating physical and psychological strategies to improve overall well-being.

Participants will be randomly assigned to one of three groups: (1) multimodal physiotherapy, (2) guided meditation via a mobile app, or (3) combined treatment. The physiotherapy program includes manual therapy, dry needling, soft tissue techniques, and cervical mobilization, delivered once a week for four weeks. The meditation program consists of daily guided sessions of approximately 5-7 minutes using the free Spanish-language content of the Insight Timer app.

Outcome measures will include pain intensity, headache-related disability, emotional state, sleep quality, mindfulness, and patient global impression of improvement, assessed at baseline, post-treatment, and at 3-month follow-up (and at 6 months if the study timeline allows).

This study aims to provide evidence for an accessible, non-invasive, and cost-effective therapeutic approach that could enhance clinical management and quality of life in people with tension-type headache.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of frequent or chronic tension-type headache (TTH) according to the International Classification of Headache Disorders, 3rd edition (ICHD-3) criteria.
* Ability to understand and communicate in Spanish sufficiently to follow instructions and complete questionnaires.
* Willingness to provide written informed consent and comply with study procedures.

Exclusion Criteria:

* Diagnosis of migraine or other primary or secondary headache disorders.
* Presence of red flags for manual therapy, including bone pathology, inflammatory disease, malignancy, neurological disorders, vestibular dysfunction, or skin infection in the cervical area.
* Fibromyalgia, pregnancy, or lactation.
* Use of pacemakers or implantable defibrillators.
* Recent medication adjustments, particularly involving psychotropic or chronic pain drugs.
* Severe psychiatric disorders (major depressive episode, bipolar disorder, schizophrenia, or other psychotic conditions).
* Previous physical treatment targeting the cranio-cervical region (manual therapy, dry needling, anesthetic blocks) within the last six months.
* Regular practice of meditation or mindfulness during the last six months.
* Participation in another clinical trial during the study period.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in headache pain intensity | Pre-allocation assessment, Baseline (Week 0), Week 4 (post-treatment), Week 12 (3-month follow-up), Week 24 (6-month follow-up)
  Headache pain intensity will be assessed using the Numerical Pain Rating Scale (NPRS, 0-10), where 0 = no pain and 10 = worst imaginable pain. Participants will record NPRS scores for each headache episode in a structured paper headache diary throughout the study (baseline, intervention, and follow-up). Weekly mean NPRS values will be calculated for statistical analysis.

SECONDARY OUTCOMES:
Change in headache frequency | Pre-allocation assessment, Baseline (Week 0), Week 4 (post-treatment), Week 12 (3-month follow-up), Week 24 (6-month follow-up)
  Number of days per week with headache, derived from the structured headache diary.
Change in mean headache duration per episode | Pre-allocation assessment, Baseline (Week 0), Week 4 (post-treatment), Week 12 (3-month follow-up), Week 24 (6-month follow-up)
  Average number of hours per headache episode, derived from the diary.
Headache Disability Inventory (HDI) | Baseline (Week 0), Week 4 (post-treatment), Week 12 (3-month follow-up), Week 24 (6-month follow-up)
  Total score and subscales (emotional and functional). Higher scores = greater disability.
Headache Impact Test (HIT-6) | Baseline (Week 0), Week 4 (post-treatment), Week 12 (3-month follow-up), Week 24 (6-month follow-up)
  Headache Impact Test (HIT-6)
Beck Depression Inventory-II (BDI-II) | Baseline (Week 0), Week 4 (post-treatment), Week 12 (3-month follow-up), Week 24 (6-month follow-up)
  Measure of depressive symptoms (0-63). Higher scores indicate greater severity.
Perceived Stress Scale-10 (PSS-10) | Baseline (Week 0), Week 4 (post-treatment), Week 12 (3-month follow-up), Week 24 (6-month follow-up)
  Scores range 0-40; higher scores = greater perceived stress.
Five Facet Mindfulness Questionnaire (FFMQ-39) | Baseline (Week 0), Week 4 (post-treatment), Week 12 (3-month follow-up), Week 24 (6-month follow-up)
  Assesses five dimensions of mindfulness; total and subscale scores analyzed.
Quality of Life (SF-36) | Baseline (Week 0), Week 4 (post-treatment), Week 12 (3-month follow-up), Week 24 (6-month follow-up)
  Eight domains scored 0-100; higher values = better perceived health.
Pittsburgh Sleep Quality Index (PSQI) | Baseline (Week 0), Week 4 (post-treatment), Week 12 (3-month follow-up), Week 24 (6-month follow-up)
  Global score 0-21; higher values = poorer sleep quality.
Insomnia Severity Index (ISI) | Baseline (Week 0), Week 4 (post-treatment), Week 12 (3-month follow-up), Week 24 (6-month follow-up)
  Global score 0-28; higher values = greater insomnia severity.

OTHER OUTCOMES:
Number of active and latent myofascial trigger points (TrPs) | Baseline (Week 0), Week 4 (post-treatment), Week 12 (3-month follow-up), Week 24 (6-month follow-up)
  The total number of active and latent myofascial trigger points will be assessed bilaterally in the upper trapezius, sternocleidomastoid, temporalis, masseter, suboccipital, and splenius capitis muscles, following international diagnostic criteria. Trigger points will be classified as active if they reproduce the participant's usual pain pattern or latent if not recognized as familiar. Examinations will be performed by an experienced physiotherapist blinded to group allocation.
Pressure Pain Thresholds (PPT) using algometry | Baseline (Week 0), Week 4 (post-treatment), Week 12 (3-month follow-up), Week 24 (6-month follow-up)
  Pressure pain thresholds will be measured bilaterally at one trigeminal point (temporal muscle), one extratrigeminal point (C5-C6 zygapophyseal joint), and two remote points (second metacarpal and tibialis anterior) using a calibrated electronic algometer. The pressure at which the sensation changes from pressure to pain will be recorded. The mean of three measurements per point will be used for analysis.
Cervical Range of Motion (CROM device) | Baseline (Week 0), Week 4 (post-treatment), Week 12 (3-month follow-up), Week 24 (6-month follow-up)
  Active cervical range of motion will be assessed using the CROM device (Performance Attainment Associates, MN, USA), which measures flexion, extension, lateral flexion, and rotation in both the global and upper cervical spine. Two measurements per movement will be taken, and the mean will be used for analysis. Assessments will be performed by a blinded physiotherapist.
Patient Global Impression of Improvement (PGI-I) | Week 4 (post-treatment), Week 12 (3-month follow-up), Week 24 (6-month follow-up)
  The PGI-I is a 7-point Likert scale that assesses the participant's perception of overall improvement, ranging from 1 = very much improved to 7 = very much worse. This measure captures the subjective evaluation of change after the intervention.
Expectation of improvement (Likert 1-10) | Baseline (Week 0)
  Before treatment begins, participants will rate their expectation of improvement using a single 10-point Likert question: "How much do you think this treatment will help your headache?" where 1 = not at all and 10 = very much. This variable will be explored as a potential covariate or predictor of treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Manuel Fernández Pérez, Pt, phD, Study Chair — Department of Physiotherapy, Faculty of Health Sciences, University of Granada; Dulce María Romero Ayuso, PhD, Study Chair — Department of Physiotherapy, Faculty of Health Sciences, University of Granada; JIHANE Boudount El Kadaoui, PT, DO, PhD(c), Study Director — Doctoral Program in Clinical Medicine and Public Health, University of Granada, Spain
Locations (1):
- J&R Global Medical Clinic S.L. (NICA 45193), Granada, Spain

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared with other researchers. All data will be anonymized and handled in accordance with the General Data Protection Regulation (EU 2016/679) and Spanish Organic Law 3/2018 on Data Protection.
  Only aggregated and de-identified results will be published in peer-reviewed journals or presented at scientific conferences.
  No transfer of raw data to third parties is planned, and data access will remain restricted to the research team at the University of Granada under the supervision of the local Biomedical Research Ethics Committee of Andalusia.

REFERENCES:
- [Background] Fernandez-de-Las-Penas C, Palacios-Cena M, Valera-Calero JA, Cuadrado ML, Guerrero-Peral A, Pareja JA, Arendt-Nielsen L, Varol U. Understanding the interaction between clinical, emotional and psychophysical outcomes underlying tension-type headache: a network analysis approach. J Neurol. 2022 Aug;269(8):4525-4534. doi: 10.1007/s00415-022-11039-5. Epub 2022 Mar 1. PMID 35229190
- [Background] Gildir S, Tuzun EH, Eroglu G, Eker L. A randomized trial of trigger point dry needling versus sham needling for chronic tension-type headache. Medicine (Baltimore). 2019 Feb;98(8):e14520. doi: 10.1097/MD.0000000000014520. PMID 30813155
- [Background] Pourahmadi M, Dommerholt J, Fernandez-de-Las-Penas C, Koes BW, Mohseni-Bandpei MA, Mansournia MA, Delavari S, Keshtkar A, Bahramian M. Dry Needling for the Treatment of Tension-Type, Cervicogenic, or Migraine Headaches: A Systematic Review and Meta-Analysis. Phys Ther. 2021 May 4;101(5):pzab068. doi: 10.1093/ptj/pzab068. PMID 33609358
- [Background] Espi-Lopez GV, Gomez-Conesa A. Efficacy of manual and manipulative therapy in the perception of pain and cervical motion in patients with tension-type headache: a randomized, controlled clinical trial. J Chiropr Med. 2014 Mar;13(1):4-13. doi: 10.1016/j.jcm.2014.01.004. PMID 24711779
- [Background] Anheyer D, Leach MJ, Klose P, Dobos G, Cramer H. Mindfulness-based stress reduction for treating chronic headache: A systematic review and meta-analysis. Cephalalgia. 2019 Apr;39(4):544-555. doi: 10.1177/0333102418781795. Epub 2018 Jun 4. PMID 29863407